CLINICAL TRIAL: NCT00526630
Title: Methylphenidate for the Treatment of Gain Impairment in Parkinson's Disease: a Randomized Double-Blind, Placebo-Controlled, Cross-over Study
Brief Title: Methylphenidate for the Treatment of Gait Impairment in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Alberto Espay, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-06-19-07
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Parkinson's Disease; Gait Impairment
Keywords: freezing; gait; festination; shuffling; balance
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. MPD (Active Comparator): Randomized to receive active Methylphenidate first. At cross-over, participants will receive placebo.
  Interventions: Drug: Methylphenidate (MPD)
- 2. Placebo (Placebo Comparator): Randomized to receive placebo first. At cross-over, participants will receive the active Methylphenidate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate (MPD) — Participants will be given 1 mg/kg of MPD divided in three doses (at 8 am, 12 noon, and 4 pm). A four-week titration period will be used, using 0.25-mg/kg increments per week until achieving the weight-adjusted target dosage, which may range from five to eight 10-mg tablets per day. The maximum daily dose will be 80 mg/day.
  Other Names: Ritalin
  Arms: 1. MPD
Drug: Placebo — Participants will be given placebo instead of active MPD.
  Arms: 2. Placebo

SUMMARY:
The purpose of this research study is to examine whether Methylphenidate (MPD) can result in improvement of gait (walking) in a population of Parkinson's Disease (PD) patients whose main disability is freezing of gait. MPD (Ritalin®) is a drug which can excite or stimulate certain systems of the body that control motor function. This drug is FDA approved for the treatment of attention hyperactivity disorder, a condition unrelated to PD.

The researchers hypothesize that daily treatment with a tolerable daily oral dose of MPD will improve gait velocity, stride length, cadence, and decrease freezing of gait, 3 months from treatment initiation in patients with moderately advanced PD, whose gait impairment is an important source of disability despite optimized antiparkinsonian treatment.

DETAILED DESCRIPTION:
There are a total of six clinic visits involved in this study. All study-related assessments will take place first during the practically defined off period, that is, in the morning after at least 12 hours from the last dose of any antiparkinsonian medication, followed by a repeat assessment once the "on" state is clearly identified by the patient and examiner (approximately 30 to 60 minutes after taking your Parkinson's medication). This "practically defined off period" state is considered the desired state on which to report motor changes for any currently available or experimental intervention in PD. Patients will be off his or her Parkinson's medication for no more than 14 hours for each of the assessments. Studying patients in the off-period is the most widely used manner in which the value of new therapies can be fully measured.

During the first visit, patients will be "randomized" into one of the study groups described below. Neither the participant nor the researcher conducting this study will choose what group he or she will be in.

Participants will receive either placebo or a dose of 1 mg/kg of Methylphenidate capsules divided into three doses (at 8 am, 12 noon, and 4 pm). An increase in medication over a four week period will be used until a target dosage is reached, which may range from 5 to 8 10-mg capsules per day.

A measure of balance will be taken during both patient's "off" and "on" motor states during each of the study visits. Patients will be asked to stand on a force plate (a piece of equipment that measures your balance and is located in the floor) for thirty seconds in a total of four conditions. The four sessions will be carried out as follows: (1) with eyes open while standing on firm surface, (2) with eyes closed while standing on firm surface, (3) with eyes open while standing on foam surface, and (4) with eyes closed while standing on foam surface. These sessions will be in random order and will be repeated up to 4 times.

During all the study visits, the physician will ask patients to perform some physical tests during which the Unified Parkinson's Disease Rating Scale (UPDRS) and the Hoehn and Yahr (H&Y) will be used to assess the severity of the patient's Parkinson's disease. Each assessment will take place during both patient's "off" and "on" motor states. Instruments that will also be used are the self-administered Freezing of Gait Questionnaire (FOGQ), to evaluate walking difficulties, and the Gait-Falls diary, to document all indoor and outdoor freezing, tripping, and falls. To assess changes in mood, patients will also complete the following instruments: the Montgomery-Asberg Depression scale (MADRS), the 15-item Geriatric Depression Scale (GDS-15) and the 20-item Zung Self-Rating Depression scale (Zung). To assess quality of life and activities of daily living, patients will complete the EQ-5D Health Questionnaire. Finally, patients will be asked to complete the Epworth Sleepiness Scale (ESS) to document any changes in sleep patterns.

After the first visit, patients will begin a four week increase in medication in order to reach a target dose. At the fourth visit, patients will receive the opposite treatment of what was received the first time and another four-week increase in medication will take place. If Methylphenidate was given at the first visit, patients will receive placebo on the third visit and vice versa. There will be a three week period where patients will not take the study medication (either Methylphenidate or placebo), between the third and fourth visit. At all study visits, during both patient's "off" and "on" motor states, patients will have balance testing. The physician will evaluate the severity of patient's disease using the UPDRS and the H&Y. Patients will be asked to complete the FOGQ and the Gait-Falls diary.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a definite diagnosis of Parkinson's disease for at least 5 years.
* Patients with mild to severe gait disturbance.
* Patients on a stable dose of anti-parkinsonian medications that will not be expected to require medication adjustments.
* Mini-Mental State Examination (MMSE) score of 25 or greater.

Exclusion Criteria:

* Patients with musculoskeletal disorders such as severe arthritis, post knee surgery, hip surgery, or any other condition that the investigators determine may impair assessment of gait.
* Previous treatment with DBS (deep brain stimulation).
* Those with history of stroke.
* Those with cerebellar, vestibular, or sensory ataxia.
* Concurrent use of, or within two weeks from discontinuing, MAO inhibitor drugs (selegiline, rasagiline).
* Women of childbearing potential.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Espay, MD, Principal Investigator — University of Cincinnati-Neurology
Locations (1):
- University Neurology-Movement Disorders Clinic, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Espay AJ, Dwivedi AK, Payne M, Gaines L, Vaughan JE, Maddux BN, Slevin JT, Gartner M, Sahay A, Revilla FJ, Duker AP, Shukla R. Methylphenidate for gait impairment in Parkinson disease: a randomized clinical trial. Neurology. 2011 Apr 5;76(14):1256-62. doi: 10.1212/WNL.0b013e3182143537. PMID 21464430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-three subjects with PD and moderate gait impairment were enrolled for this 6-month placebo-controlled, double-blind study.
Groups:
- MPD Then Placebo: First group treated with MPD then placebo
- Placebo Then MPD: First group treated with placebo then MPD
Period: First Intervention Period - 12 Weeks
Arm/Group | MPD Then Placebo | Placebo Then MPD
Started | 12 | 11
Completed | 12 | 8
Not Completed | 0 | 3
Not completed — Withdrawn | 0 | 3
Period: Second Intervention Period - 12 Weeks
Arm/Group | MPD Then Placebo | Placebo Then MPD
Started | 12 | 8
Completed | 10 | 7
Not Completed | 2 | 1
Not completed — Withdrawn | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were randomized to receive both MPD and placebo.
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Secondary Outcome: The Unified Parkinson Disease Rating Scale (UPDRS) Between Groups at 12 and 27 Weeks
Description: Patients will have a mild to severe gait disturbance with score >1 on the motor subscale of the Unified Parkinson's disease rating scale (UPDRS) but without need for a continuous ambulatory aid such as walker or wheelchair (Hoehn & Yahr 2-3). The highest score possible for the UPDRS is 108 which indicates severe motor impairment. The lowest score for the UPDRS is 0 which indicates no motor impairment.
Time Frame: At week 12 and 27
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Baseline gait composite scores
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
units on a scale | 21.18 (12.73) | 20.33 (10.48) | 18.39 (8.21)

2. Primary Outcome: The Primary Outcome Measure Was Change in a Gait Stride Length Between Groups at 12 and 27 Weeks.
Description: Gait stride length is the distance between two consecutive steps in the "on" state. This will be measured by the GAITRite System, which is an electronic walkway utilized to measure the temporal (timing) and spatial (two dimension geometric position) parameters of its pressure activated sensors.
Time Frame: Week 12 and 27
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Baseline: All participants with baseline data
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
centimeters | 107.66 (26.03) | 112.29 (21.85) | 103.35 (24.24)

3. Primary Outcome: The Primary Outcome Measure Was Change in Gait Velocity Between Groups at 12 and 27 Weeks.
Description: Gait velocity is a measure of distance over time in the "on" state. This will be measured by the GAITRite System, which is an electronic walkway utilized to measure the temporal (timing) and spatial (two dimension geometric position) parameters of its pressure activated sensors.
Time Frame: Week 12 and 27
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
centimeters/second | 96.96 (22.38) | 99.24 (15.16) | 95.76 (25.38)

4. Secondary Outcome: Duration of Freezing and Shuffling Episodes Between Groups at 12 and 27 Weeks.
Description: Freezing and shuffling are measures of ambulatory impairment.
Time Frame: Week 12 and 27
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
hours
  Shuffling | 7.67 (5.02) | 6.15 (4.05) | 9.1 (3.7)
  Freezing | 3.07 (2.99) | 3.25 (3.02) | 5.4 (4.11)

5. Secondary Outcome: Freezing of Gait Questionnaire (FOGQ) Scores Between Groups at 12 and 27 Weeks.
Description: FOGQ is a questionnaire that quantifies severity of gait and falls. It contains 16 items with a 0-4 severity scale for each, for a range of 0 (normal) to 64 (most severe impairment).
Time Frame: Week 12 and 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
units on a scale | 12.31 (2.73) | 12.56 (4.11) | 12.71 (3.87)

6. Secondary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS) Between Groups at 12 and 27 Weeks.
Description: MADRS is a questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60
Time Frame: Week 12 and 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
units on a scale | 5.79 (5.24) | 6.71 (6.2) | 9.44 (5.93)

7. Secondary Outcome: The Epworth Sleepiness Scale (ESS) Between Groups at 12 and 27 Weeks
Description: The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness that is measured by use of a very short questionnaire. The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, though not necessarily every day. The scores for the eight questions are added together to obtain a single number. A number in the 0-9 range is considered to be normal while a number in the 10-24 range indicates excessive daytime sleepiness. Higher scores imply worse sleepiness.
Time Frame: Week 12 and 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
units on a scale | 11.05 (4.55) | 10.71 (3.7) | 11.24 (3.53)

8. Secondary Outcome: The 5-item EuroQoL (EQ-5D) Quality of Life Generic Instrument Between Groups at 12 and 27 Weeks.
Description: The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem; see appendix). A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The range is from 0 to 100, with 100 indicating the best health status.
Time Frame: Week 12 and 27
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1. MPD | 2. Placebo | Baseline
Number analyzed (Participants) | 20 | 23 | 23
units on a scale | 65 (25.7) | 63.94 (20.71) | 68.67 (13.56)

ADVERSE EVENTS:
Time Frame: Adverse event data was captured during the course of the study either by phone interview or at the study visit.
Arm/Group | 1. MPD | 2. Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 5/20 | 5/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. MPD (N=20) | 2. Placebo (N=23)
irritability (Psychiatric disorders) | 5 (5) | 0 (0)
Loss of bladder control (Renal and urinary disorders) | 1 | 0
Double vision (Eye disorders) | 1 | 0
Bad nightmares, transient (Nervous system disorders) | 1 | 0
Less dyskinesia (Nervous system disorders) | 1 | 1
More dyskinesia (Nervous system disorders) | 3 | 1
Sleep improved (Nervous system disorders) | 2 | 1
Sleep deteriorated (Nervous system disorders) | 2 | 0
No strength or energy (Nervous system disorders) | 5 | 1
Stiffness, soreness, cramps (Nervous system disorders) | 2 | 2
Visual hallucinations (Nervous system disorders) | 2 | 1
Crying (General disorders) | 1 | 0
Suppressed appetite (Gastrointestinal disorders) | 2 | 1
Lightheadedness (Nervous system disorders) | 1 | 0
Increased wakefulness (Nervous system disorders) | 1 | 0
Decreased soreness (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 1
Confusion, forgetfulness (Nervous system disorders) | 0 | 4
Flushing (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No